CLINICAL TRIAL: NCT01944644
Title: The Effect of Low Field Magnetic Stimulation on Resting State Networks in Major Depressive Disorder
Brief Title: Low Field Magnetic Stimulation for Treatment Resistant Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1207012777; 1207012777 (Other: Weill Cornell Medical College IRB)
Record Dates: First submitted 2013-09-12; First posted 2013-09-17 (Estimated); Results first posted 2018-09-17 (Actual); Last update posted 2018-09-17 (Actual); Status verified 2018-08

CONDITIONS: Treatment Resistant Depression
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Active Low Field Magnetic Stimulation (Active Comparator): LFMS will follow a previously published protocol for the treatment of a Major Depressive Episode (Rohan et al. 2004). Active Low Field Magnetic Stimulation treatments will be delivered with a prototype LFMS device manufactured by Tal Medical. LFMS sessions consist of proton echo-planar magnetic resonance spectroscopic imaging (EP-MRSI) and will be 20min in duration. LFMS exposes subjects to magnetic fields of the same magnitude and frequency used in clinical MR-Spectroscopic imaging of the brain.
  Interventions: Device: Active Low Field Magnetic Stimulation
- Sham Low Field Magnetic Stimulation (Sham Comparator): Sham Low Field Magnetic Stimulation will consist of a three-dimensional spoiled gradient echo sequence of the same duration as active LFMS and which provides auditory stimulation indistinguishable from active treatment.
  Interventions: Device: Sham Low Field Magnetic Stimulation

INTERVENTIONS:
Device: Active Low Field Magnetic Stimulation — Active Low Field Magnetic Stimulation treatments will be delivered with a prototype LFMS device manufactured by Tal Medical. LFMS sessions consist of proton echo-planar magnetic resonance spectroscopic imaging (EP-MRSI) and will be 20min in duration. LFMS exposes subjects to magnetic fields of the same magnitude and frequency used in clinical MR-Spectroscopic imaging of the brain.
  Arms: Active Low Field Magnetic Stimulation
Device: Sham Low Field Magnetic Stimulation — Sham Low Field Magnetic Stimulation will consist of a three-dimensional spoiled gradient echo sequence of the same duration as active LFMS and which provides auditory stimulation indistinguishable from active treatment.
  Arms: Sham Low Field Magnetic Stimulation

SUMMARY:
This is a double-blind, randomized, sham-controlled phase II study of the effects of Low Field Magnetic Stimulation (LFMS) on brain circuitry of adults with treatment-resistant Major Depressive Disorder (MDD). Eligible subjects will be randomly assigned to double-blind treatment with three 20 minute sessions of either (1) active LFMS or (2) sham LFMS. Resting state fMRI will be performed at baseline and following the third and final treatment session.

DETAILED DESCRIPTION:
A minimum of 60 subjects will enter the double-blind treatment phase of the study. This trial will be conducted according to the U.S. Food and Drug Administration guidelines and the Declaration of Helsinki. Written informed consent will be obtained from all patients before protocol-specified procedures are carried out. The subjects will be drawn from an outpatient sample of patients with current Major Depressive Disorder (MDD) diagnosed with the use of the Mini International Neuropsychiatric Interview (MINI).

LFMS will follow a previously published protocol for the treatment of a Major Depressive Episode (Rohan et al. 2004). LFMS treatments will be delivered with a prototype LFMS device manufactured by Tal Medical. LFMS sessions consist of proton echo-planar magnetic resonance spectroscopic imaging (EP-MRSI) and will be 20min in duration. LFMS exposes subjects to magnetic fields of the same magnitude and frequency used in clinical MR-Spectroscopic imaging of the brain. Sham LFMS will consist of a three-dimensional spoiled gradient echo sequence of the same duration as active LFMS and which provides auditory stimulation indistinguishable from active treatment.

At the beginning of a treatment session, the subject will sit in front of and position his head within the open bore of the Tal Medical LFMS device. The device will be pre-programmed to deliver active or sham treatment so that the subject, operator, and all investigators are blinded to active treatment vs. sham. Immediately before and after each treatment session, the PANAS, Ham-D-6, and Visual Analog Mood Scale will be administered and the patient will be monitored for any adverse events.

All participants will undergo two sessions of neuroimaging: On the Friday prior to the first treatment session (Day 0) and on the day of the third and final treatment session (Day 7). Each session of neuroimaging will be 50 minutes in duration and include three imaging modalities: Resting State fMRI (rsfMRI), Arterial Spin Labeling MRI (ASL), and Diffusion Tensor Imaging (DTI). In addition, we will obtain high-resolution anatomical volumes (SPGR) for each subject for the purpose of transforming each individual's imaging data into a common space for group comparisons. Subjects will lie still in the scanner and will be instructed to let their mind "wander freely" during the acquisition of the resting state fMRI scan, which will last 6 minutes (Anon 2001). They will also be instructed to lie still during the ASL and DTI scans (each lasting 8 minutes). In addition, we will obtain a high-resolution T1-weighted (MP-RAGE) anatomical scan for co-registration of each individual's imaging data into a common space for group statistics..

Resting state fMRI will be used to measure the functional connectivity within the default mode network (DMN) and other circuits that are known to function abnormally in MDD (Greicius et al. 2007). ASL will be used to measure the regional blood flow within individual nodes of this circuitry, while DTI will measure the structural integrity of the connections between nodes. Measurements at baseline will be compared to measurements post-LFMS in both active treatment and sham groups.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be able to understand and read English and give written informed consent prior to the protocol required procedures.
2. Men and women, ages 18 to 65 inclusive with a diagnosis of major depressive episode as defined by DSM-IV-TR criteria.
3. History of an inadequate response to 1 or more adequate antidepressant treatments in the current depressive episode.
4. Subjects must have a 17-item Hamilton Rating Scale for Depression (HAM-D-17) score ≥ 18.
5. Subjects must have a Body Mass Index (BMI) of approximately 18-40 kg/m².
6. Women of childbearing potential (WOCBP) must be using an adequate method of contraception to avoid pregnancy throughout the study and must have a negative urine pregnancy test within 72 hours prior to the start of LFMS.

Exclusion Criteria:

1. WOCBP who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period.
2. Women who are pregnant or breastfeeding.
3. Subjects with other DSM-IV-TR Axis I disorders other than Generalized Anxiety Disorder (GAD: 300.02), Social Anxiety Disorder (300.23), or Specific Phobia (300.29). Subjects with co-morbid GAD, Social Anxiety Disorder, or Specific Phobia are ineligible if the co-morbid condition is clinically unstable, requires treatment, or has been the primary focus of treatment within the 6 month period prior to screening.
4. Delirium, dementia, or other cognitive disorder
5. Schizophrenia or other psychotic disorder, based on the MINI.
6. Patients with a clinically significant Axis II diagnosis of borderline, antisocial, paranoid, schizoid, schizotypal or histrionic personality disorder.
7. Patients experiencing hallucinations, delusions, or any psychotic symptomatology in the current or any previous depressive episode.
8. Patients who have met DSM-IV-TR criteria for any significant substance use disorder within the past six months.
9. Patients receiving new-onset psychotherapy and/or somatic therapy (light therapy, transcranial magnetic stimulation) within 6 weeks of screening, or at any time during participation in the trial.
10. Patients who, in the opinion of the Investigator, are actively suicidal and at significant risk for suicide.
11. Patients who have participated in any clinical trial with an investigational drug or device within the past month.
12. Patients who have received ECT in the past 20 years or Vagal Nerve/Deep Brain Stimulation during their lifetime.
13. Unstable medical illness including, cardiovascular, hepatic, renal, respiratory, endocrine, neurological, or hematological disease.
14. Subjects with evidence or history of significant neurological disorder, including head trauma with loss of consciousness, history of stroke, Parkinson's disease, epilepsy disorder, conditions that lower seizure threshold, seizures of any etiology (including substance or drug withdrawal), who are taking medications to control seizures, or who have increased risk of seizures as evidenced by history of EEG with epileptiform activity (with the exception of juvenile febrile seizures).
15. Patients with thyroid pathology (unless condition has been stabilized with medications for at least the past three months).
16. Patients who have recently (within two weeks) begun any medications.
17. Monoamine oxidase inhibitors (e.g., Nardil, phenelzine, Parnate, tranylcypromine, Marplan, isocarboxazide) treatment within the 2 weeks prior to enrollment.
18. Patients with a history of antidepressant-induced hypomania or dysphoria.
19. Participants with metal implants (Will use the NY Presbyterian Hospital MRI Checklist)
20. Any of the following exclusion criteria for MRI Cardiac pacemaker or pacing wires Implanted cardioverter defibrillator (ICD) Cochlear, otologic, or other ear implant Tissue expander (e.g., breast) Implanted drug infusion device Aneurysm clip(s) Deep Brain Stimulator Other Neuro-stimulator Prosthesis (eye, penile, limb, etc.) Artificial heart valve Eyelid spring or wire Stent, filter, or coil Programmable shunt Catheter or feeding tube with metal tip Radiation seeds Medication patch (Nicotine, Nitroglycerine) Any metallic fragment, foreign body or bullets Surgical staples, clips, metallic sutures or wire mesh Bone/joint pin, screw, nail, wire, plate, etc. IUD, diaphragm, or pessary Dentures or braces Tattoo, permanent makeup or body piercing jewelry Hearing aid (Remove before entering the MR system room) Breathing problem and motion disorder Claustrophobia Hair Extensions

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2013-08; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc Dubin, MD, PhD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Participants will be able to find out which treatment arm they were assigned at the conclusion of the study.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active Low Field Magnetic Stimulation | Sham Low Field Magnetic Stimulation
Started | 34 | 32
Completed | 34 | 32
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Low Field Magnetic Stimulation | Sham Low Field Magnetic Stimulation | Total
Number analyzed (Participants) | 34 | 32 | 66
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.6 (15.1) | 46.2 (12.2) | 46.4 (13.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 20 | 37
  Male | 17 | 12 | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 5 | 9
  Not Hispanic or Latino | 30 | 27 | 57
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 8 | 15
  White | 26 | 22 | 48
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 34 | 32 | 66
Hamilton Scale for Depression (HamD) 6 Item [Mean (Standard Deviation); unit: units on a scale] — The Hamilton Scale for Depression 6 item subscale scores range from 0-24. Higher scores indicate greater severity of depression. Total scores are reported with no subscales.
  units on a scale | 11.8 (1.7) | 11.4 (1.8) | 11.6 (1.75)
Visual Analog Scale [Mean (Standard Deviation); unit: units on a scale] — A Visual Analog Scale is a measurement of subjective characteristics that cannot be directly measured. Using this self questionnaire, subjects specify their level of depression along a continuous line between two end-points ranging from 0-100 (higher score means better mood).
  units on a scale | 55.4 (19.9) | 49.9 (21.8) | 52.7 (20.1)
Positive and Negative Affect Score (PANAS) - Negative Subscale [Mean (Standard Deviation); unit: units on a scale] — The Positive and Negative Affect Schedule (PANAS) measures both positive affect and negative affect. Participants in the PANAS are required to respond to two 20-item subscales using 5-point scale that ranges from very slightly or not at all (1) to extremely (5). This negative subscale captures self-rated scale of symptoms of depression ranging from 0-50 (higher score means worse depression).
  units on a scale | 23.7 (7.6) | 27.5 (8.9) | 25.6 (8.25)
Positive and Negative Affect Score (PANAS) - Positive Subscale [Mean (Standard Deviation); unit: units on a scale] — The Positive and Negative Affect Schedule (PANAS) measures both positive affect and negative affect. Participants in the PANAS are required to respond to two 20-item subscales using 5-point scale that ranges from very slightly or not at all (1) to extremely (5). This positive subscale captures self-rated scale of symptoms of depression ranging from 0-50 (higher score means less depression).
  units on a scale | 23.1 (8.7) | 22.4 (8.0) | 22.8 (8.4)

OUTCOME MEASURES:

1. Primary Outcome: 6 Item Hamilton Depression Rating Scale
Description: This is to compare the 6 Item Hamilton Depression Rating Scale from the Screen to after 3 Sessions of Active or Sham LFMS (7 days post-baseline). The Hamilton Scale for Depression 6 item subscale scores range from 0-24. Higher scores indicate greater severity of depression. Total scores are reported with no subscales.
Time Frame: 7 days after baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active Low Field Magnetic Stimulation | Sham Low Field Magnetic Stimulation
Number analyzed (Participants) | 34 | 32
units on a scale | 7.4 (3.4) | 7.6 (3.7)

2. Primary Outcome: Visual Analog Scale
Description: A Visual Analog Scale is a measurement of subjective characteristics that cannot be directly measured. Using this self questionnaire, subjects specify their level of depression along a continuous line between two end-points ranging from 0-100 (higher score means better mood).
Time Frame: 7 days after baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active Low Field Magnetic Stimulation | Sham Low Field Magnetic Stimulation
Number analyzed (Participants) | 34 | 32
units on a scale | 74 (20.6) | 59.4 (26.2)

3. Primary Outcome: Positive and Negative Affect Score (PANAS) - Negative Subscale
Description: The Positive and Negative Affect Schedule (PANAS) measures both positive affect and negative affect. Participants in the PANAS are required to respond to two 20-item subscales using 5-point scale that ranges from very slightly or not at all (1) to extremely (5). This negative subscale captures self-rated scale of symptoms of depression ranging from 0-50 (higher score means worse depression).
Time Frame: 7 days after baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active Low Field Magnetic Stimulation | Sham Low Field Magnetic Stimulation
Number analyzed (Participants) | 34 | 32
units on a scale | 15.8 (7.2) | 18.6 (7.4)

4. Primary Outcome: Positive and Negative Affect Score (PANAS) - Positive Subscale
Description: The Positive and Negative Affect Schedule (PANAS) measures both positive affect and negative affect. Participants in the PANAS are required to respond to two 20-item subscales using 5-point scale that ranges from very slightly or not at all (1) to extremely (5). This positive subscale captures self-rated scale of symptoms of depression ranging from 0-50 (higher score means worse depression).
Time Frame: 7 days after baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active Low Field Magnetic Stimulation | Sham Low Field Magnetic Stimulation
Number analyzed (Participants) | 34 | 32
units on a scale | 24.8 (8.7) | 25.5 (11.9)

ADVERSE EVENTS:
Time Frame: 7 days.
Arm/Group | Active Low Field Magnetic Stimulation | Sham Low Field Magnetic Stimulation
All-Cause Mortality (participants affected / at risk) | 1/34 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/32
Other Adverse Events (participants affected / at risk) | 1/34 | 0/32
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Low Field Magnetic Stimulation (N=34) | Sham Low Field Magnetic Stimulation (N=32)
Panic Attack (Psychiatric disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes